CLINICAL TRIAL: NCT05459740
Title: The Relations of Resilience to Self-management Behaviors Among Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Self-management Behaviors and Resilience Among Chronic Obstructive Pulmonary Disease Patients
Status: Completed | Type: Observational
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20191101R
Record Dates: First submitted 2022-06-27; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Self-management Behavior; Resilience
Keywords: chronic obstructive pulmonary disease; self-management behavior; resilience
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study conducted an assessment of the influencing factors and correlations that affect self-management behaviors and resilience in the COPD population.

DETAILED DESCRIPTION:
A total of 100 participants with COPD from a medical center in Northern Taiwan were recruited from February 2020 to January 2021 in this cross-sectional study. Each subject completed self-reported questionnaires through face-to-face interviews, including 20-item COPD Self-Management Scale (CSMS-20) and a 25-item Connor-Davidson Resilience Scale (CD-RISC-25). A multiple linear regression model was used to examine the relationship between the levels of self-management behavior and resilience, controlling for sociodemographic and clinical factors.

ELIGIBILITY:
Inclusion Criteria:

The recruited participants have been diagnosed with COPD for at least a month by thoracic physicians based on the guidelines of the Global Initiative for Chronic Obstructive Lung Disease (GOLD).

Exclusion Criteria:

Participants who were diagnosed with serious mental disorders, cancer, terminal illness, or end-stage diseases were excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The age ranged from 39-90 years old for all the population. The proportions of BMI < 18.5 kg/m2, 18.5-24.9 kg/m2, and ≥ 24.9 kg/m2 were 8%, 58%, and 34%, respectively. Overall, only 14% of the COPD subjects were educated with a university degree or higher, which was associated with higher self-management scores compared to those educated with below university degree. Half of the subjects were former smokers.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Levels of COPD self-management behavior | 2020-02-01 to 2021-01-30
  Each subject completed the self-reported 20-item COPD Self-Management Scale (CSMS-20) questionnaire through face-to-face interviews. The range of scores is from 20 to 100, with a higher score indicating better self-management behaviors.
Levels of COPD psychological resilience | 2020-02-01 to 2021-01-30
  Each subject completed the 25-item Connor-Davidson Resilience Scale (CD-RISC-25) questionnaire through face-to-face interviews. The range of scores is from 0 to 100, with a higher score indicating better psychological resilience.

CONTACTS AND LOCATIONS:
Overall Officials: EN-MING CHANG, master, Study Chair — Respiratory therapist
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No